CLINICAL TRIAL: NCT00549926
Title: Yokohama Assessment of Fluvastatin, Pravastatin, Pitavastatin and Atorvastatin in Acute Coronary Syndrome (Yokohama-ACS)
Acronym: Yokohama-ACS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yokohama City University Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Yokohama-ACS
Record Dates: First submitted 2007-10-25; First posted 2007-10-26 (Estimated); Last update posted 2010-02-17 (Estimated); Status verified 2010-02

CONDITIONS: Coronary Disease; Hypercholesterolemia
MeSH Terms: conditions — Coronary Disease; Hypercholesterolemia | interventions — Fluvastatin; Pravastatin; pitavastatin; Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Active Comparator)
  Interventions: Drug: Fluvastatin
- 2 (Active Comparator)
  Interventions: Drug: Pravastatin
- 3 (Active Comparator)
  Interventions: Drug: Pitavastatin
- 4 (Active Comparator)
  Interventions: Drug: Atorvastatin

INTERVENTIONS:
Drug: Fluvastatin
  Arms: 1
Drug: Pravastatin
  Arms: 2
Drug: Pitavastatin
  Arms: 3
Drug: Atorvastatin
  Arms: 4

SUMMARY:
The purpose of this study is to compare the effects of fluvastatin, pravastatin, pitavastatin, and atorvastatin on coronary plaque volume in patients with acute coronary syndrome, and to clarify the impact of moderate and intensive lipid lowering therapy on coronary plaque volume, serum lipids, and inflammation markers in patients with acute coronary syndrome in Japanese.

DETAILED DESCRIPTION:
Previous mega trials have demonstrated that lipid lowering therapy with HMG-CoA reductase inhibitors (statins) reduces the incidence of major cardiovascular events by one-third, thus, the benefit of lipid lowering therapy has been substantiated. Such a benefit is significant especially for patients with coronary heart disease (CHD). The third report of the National Cholesterol Education Program Adult Treatment Panel (NCEP ATP-III) has suggested the advantage of more intensive lipid lowering therapy with a goal of reducing LDL-C below 70 mg/dL for such patients categorized as very high risk. In Japan, Japan Atherosclerosis Society (JAS) Guidelines for Diagnosis and Treatment of Atherosclerotic Cardiovascular Diseases 2002 have recommended that an LDL-C goal for patients with coronary heart disease should be below 100 mg/dL. However, there is no satisfactory evidence whether we need to lower LDL-C level less than the 70mg/dL or not in Japanese population.

Recently, research on diagnosis of coronary plaque has shown significant advances. The REVERSAL study in patients with a history of CHD, by diagnosis with intravascular ultrasound, suggested that intensive lipid lowering therapy with atorvastatin (80 mg/day) was associated with no growth of plaque (-0.4% compared to baseline), whereas therapy with pravastatin (40 mg/day) showed a slight increase (2.7%) in plaque volume over 18 months in Western population.

In Japanese population, MEGA study have shown the effect of moderate lipid lowering therapy in primary prevention of cardiovascular events. However, the effect of moderate lipid lowering therapy in secondary prevention of cardiovascular events is unknown.

Pravastatin and fluvastatin are the statin which has been administered in Japan for several years.

Although LDL-C lowering effect of these statins were less strong than new generation statins, their safeｔｙ profile have been well established. Fluvastatin were expected to reduce coronary plaque because of its high affinity to arterial tissue and antioxygenic effect compared with pitavastatin, but the effect on human coronary plaque has not been reported.

Relative plaque regression rate between intensive and moderate lipid lowering therapy would clarify the ideal level of target LDL-C in Japanese population. Furthermore, the different effect on coronary plaque between pravastatin and fluvastatin which have similar LDL-C lowering effect and different affinity to arterial tissue would determine the superior lipid lowering regimen to affect coronary plaque volume.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who have been diagnosed as acute coronary syndrome, and successful percutaneous coronary intervention (PCI) were performed with intravascular ultrasound (IVUS) guidance.
2. Patients having coronary plaques (≧ 500 µm in thickness or % plaque of 20% or more at ≧ 5 mm distal or proximal to the previously treated area in the same branch of coronary artery.
3. Patients with hypercholesterolemia as defined by any of the following criteria:

   * TC ≧ 220 mg/dL
   * LDL-C ≧ 140 mg/dL Cholesterol-lowering treatment is allowed according to the investigator's judgement when LDL-C ≧ 100 mg/dL or TC ≧ 180 mg/dL.
4. Patients with written consent by their own volition after being provided sufficient explanation for their participation in this clinical trial.
5. Patients 20 years or older at the time of their consent.

Exclusion Criteria:

1. Patients with bypass graft or in-stent restenosis at the site of PCI.
2. Patients who received PCI in the past on the lesion where the evaluation of coronary plaque volume is planned.
3. Patients who had plaques in a non-culprit site and might receive PCI during the treatment period.
4. Patients receiving lipid-lowering drugs (statins, fibrates, probucol, nicotinic acid or cholesterol absorption inhibitors).
5. Patients with familial hypercholesterolemia.
6. Patients with cardiogenic shock.
7. Patients receiving cyclosporine.
8. Patients with any allergy to pravastatin, fluvastatin, pitavastatin, or atorvastatin.
9. Patients with hepatobiliary disorders.
10. Pregnant women, women suspected of being pregnant, or lactating women.
11. Patients with renal disorders or undergoing dialysis.
12. Patients who are ineligible in the opinion of the investigator.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2007-10; Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
the percent change in coronary plaque volume the percent change in integrated backscatter signal obtained by integrated backscatter IVUS | 9-11 month

SECONDARY OUTCOMES:
absolute change from baseline in coronary plaque volume | 9-11 month
absolute and percent changes in minimal lumen diameter(MLD) and percent(%) stenosis | 9-11 month
absolute and percent changes in total cholesterol(TC);low-density lipoprotein(LDL)-cholesterol(LDL-C) | 9-11 month

CONTACTS AND LOCATIONS:
Overall Officials: Naohiro Komura, Principal Investigator — Yokohama City University Medical Center
Locations (1):
- Yokohama City University Medical Center, Yokohama, Japan

REFERENCES:
- [Derived] Matsushita K, Hibi K, Komura N, Kimura Y, Matsuzawa Y, Konishi M, Maejima N, Iwahashi N, Kosuge M, Ebina T, Tamura K, Kimura K. Impact of serum lipoprotein (a) level on coronary plaque progression and cardiovascular events in statin-treated patients with acute coronary syndrome: a yokohama-acs substudy. J Cardiol. 2020 Jul;76(1):66-72. doi: 10.1016/j.jjcc.2020.01.005. Epub 2020 Feb 7. PMID 32037254
- [Derived] Hibi K, Sonoda S, Kawasaki M, Otsuji Y, Murohara T, Ishii H, Sato K, Koshida R, Ozaki Y, Sata M, Morino Y, Miyamoto T, Amano T, Morita S, Kozuma K, Kimura K, Fujiwara H; Ezetimibe-ACS Investigators. Effects of Ezetimibe-Statin Combination Therapy on Coronary Atherosclerosis in Acute Coronary Syndrome. Circ J. 2018 Feb 23;82(3):757-766. doi: 10.1253/circj.CJ-17-0598. Epub 2017 Dec 7. PMID 29212965